CLINICAL TRIAL: NCT03737513
Title: Exercise-induced Collective Rhabdomyolysis
Status: Completed | Type: Observational
Sponsor: Haitao Tu (Other)
Collaborators: Yueqing Hospital Affiliated to Wenzhou Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Haitao Tu, Attending physician, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Organization: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Other Study IDs: 2018110801
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Rhabdomyolysis
Keywords: Rhabdomyolysis; Military Training
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — whole blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rhabdomyolysis, which is a characteristic occurrence in associated with muscle cell necrosis, develops due to various causes.The investigators herein report a rare case of collective rhabdomyolysis after high intensity resistance training, including 35 teenagers（participants），in which markedly elevated levels of serum creatine kinase (CK) and serum myoglobin were observed. This high intensity resistance trainings is a part of Military Training(MT)，which all the middle school students must finish before admission。

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rhabdomyolysis;
* Caused by military training;
* Informed consent；
* Must be able to cooperate with blood test.

Exclusion Criteria:

* Caused by drugs and other reasons;
* No hospitalization event

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Students who participated in this military training from the same school
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
serum creatine kinase； | 3 months
  Change in serum creatine kinase at 3 months
serum myoglobin | 1 week
  At the time of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Yueqing Hospital Affiliated to Wenzhou Medical University, Yueqing, Zhejiang, China